CLINICAL TRIAL: NCT04914260
Title: Injured - Sport Health Armed Forces (Blessé - Sport Santé Armées): Reconstruction Through Sport in the Armed Forces
Acronym: B-SSA
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PPRC25; 2021-A00718-33 (Other: IDRCB)
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Physical Injury
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — The participants will have to fill in an on-line questionnaire regarding quality of life, their level of knowledge of the rehabilitation through sport program and their level of satisfaction toward this program.

SUMMARY:
Since 2014, the armed forces have been offering injured military personnel the opportunity to rebuild their lives through sport. Sport, considered as the "DNA" of the military, thus becomes a vector of socio-professional reintegration for physically and psychologically injured soldiers.

In its 2019-2024 national Sport-Health strategy and in the Ministry of the Armed Forces' "Sport 2025" plan, rebuilding injured military personnel through sport is becoming a major focus of the new sports policy for the armed forces.

In addition to the well identified physiological benefits, sports are recognized as a way to encourage social relationships, fight stress and isolation, and promote solidarity. Sport thus contributes to the physical and mental reconstruction of the injured, promoting the phenomenon of resilience well described in the Anglo-Saxon world.

The implementation of the Reconstruction through Sport Program ("PRS") is based on the coordinated actions of the assistance units for the wounded, the French Armed Forces Health Service and the National Center for Defense Sports (CNSD), which have set up a complete sports program (discovery, leisure, competitions), adapted and evolving, regardless of the physical and/or psychological after-effects and the disability secondary to the injury.

In France, there are an increasing number of PRS-labeled sports events, such as the Military Injury and Sports Meetings, the Ad Victoriam Challenge, and internationally, the Invictus Games and the Military World Games. It should also be noted that this pathway leads some injured people to high-level competition.

No study has yet evaluated the path of reconstruction through sport for French injured military personnel initiated in 2014.

ELIGIBILITY:
Inclusion Criteria:

* French military
* Physically injured since January 1st, 2008
* Registered by a casualty assistance cell
* On duty or on long term sick leave

Exclusion Criteria:

* No physical injury
* Individuals who do not speak, understand or read French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of French soldiers who have been physically injured and have been registered by a casualty assistance cell.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Level of knowledge of the rehabilitation through sport program | At enrollment
  The level of knowledge will be assessed through 3 questions scored from 0 (absence of knowledge) to 10 (perfect knowledge).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'Instruction des Armées Percy, Clamart, France

IPD SHARING:
Plan to Share IPD: Undecided